CLINICAL TRIAL: NCT02024854
Title: Skin-to-skin After Delivery in Preterm Infants Born at 28-32 Weeks of Gestation. A Randomized Controlled Trial
Brief Title: Skin-to-skin After Delivery in Preterm Infants Born at 28-32 Weeks of Gestation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Drammen sykehus (Other); Sorlandet Hospital HF (Other Government); IWK Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KC28-32
Record Dates: First submitted 2013-12-19; First posted 2013-12-31 (Estimated); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Premature Birth
Keywords: Kangaroo-Mother Care Method; Stress, Physiological
MeSH Terms: conditions — Premature Birth | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- skin-to-skin (Experimental): immediately after birth the baby is laid on mother's chest for as long as justifiable medically to max 2 hours.
  Interventions: Behavioral: skin-to-skin
- standard care (Active Comparator): after birth the baby is transferred to the neonatal intensive care unit
  Interventions: Behavioral: standard care

INTERVENTIONS:
Behavioral: skin-to-skin
  Arms: skin-to-skin
Behavioral: standard care
  Arms: standard care

SUMMARY:
The aim of the study is to investigate physiological response, social/emotional response and general movements in preterm infants when they are given skin-to-skin contact with the mother (intervention) or standard care (incubator) right after delivery. Preterm infants will be randomized to either intervention or standard care group. Data on body temperature, blood glucose, hart rate, respiration rate and oxygen saturation will be obtained. In addition the infant will be video-recorded during the first 24 hours and at three months of age for analysis of the general movements.

DETAILED DESCRIPTION:
Power calculations are based on a difference in Bayley Scale of Infant Development III, cognitive scale at two years corrected age of about 7,5 mean score =0.5 SD (α=0,05, β=0.80). Based on this analysis, 64 preterm infants are needed in each group to yield statistic significance. Allowing for withdrawals, the sample size is set to 68 in each group.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants at 28-32 weeks of gestation (born 12-8 weeks before term)

Exclusion Criteria:

* Infants who need immediate medical interventions

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
cognitive scorer at two years corrected age | 2 year
  measured by Bayley Scales of Infant Development Third Edition (BSID III)

SECONDARY OUTCOMES:
change in heart rate | 24 hours
change in body temperature | 24 hours
change in respiration frequency | 24 hours
change in blood glucose | 24 hours
general movements (GM) at 3 months corrected age | 3 months
  assessed with the General Movement Assessment (GMA)
Nutrition | 1 year
  based on a Norwegian questionnaire, based on a Norwegian national survey from The Norwegian Directorate of Health.
Social/emotional competence at three months corrected age | 3 months
  measured with the Ages and Stages Questionnaire: Social Emotional (ASQ:SE)
Social/emotional competence at two years corrected age | 1 year
  measured with the Ages and Stages Questionnaire: Social Emotional (ASQ:SE)
Social/emotional competence at two years corrected age | 2 years
  measured with the Ages and Stages Questionnaire: Social Emotional (ASQ:SE)
Developmental skills at two years corrected age | 1 year
  measured with the Ages and Stages Questionnaire: (ASQ)
Developmental skills at two years corrected age | 2 years
  measured with the Ages and Stages Questionnaire: (ASQ)
Maternal anxiety | at discharge from hospital
  measured with State-Trait Anxiety Inventory (STAI)
Maternal anxiety | 3 months
  measured with State-Trait Anxiety Inventory (STAI)
Maternal anxiety | 2 years
  measured with State-Trait Anxiety Inventory (STAI)
Child Behaviour | 5 year
  Measured with Child Behaviour Checklist

CONTACTS AND LOCATIONS:
Overall Officials: Håkon Bergseng, md phd, Study Director — Norwegian University of Science and Technology
Locations (4):
- IWK Health Centre, Halifax, Canada
- Norway (3):
  - Nyfødt intensiv, Drammen sykehus, Drammen
  - Nyfødt intensiv, Sørlandet Sykehus, Kristiansand
  - NICU St Olavs Hospital, Trondheim

REFERENCES:
- [Background] Kristoffersen L, Stoen R, Rygh H, Sognnaes M, Follestad T, Mohn HS, Nissen I, Bergseng H. Early skin-to-skin contact or incubator for very preterm infants: study protocol for a randomized controlled trial. Trials. 2016 Dec 12;17(1):593. doi: 10.1186/s13063-016-1730-5. PMID 27955652
- [Derived] Kristoffersen L, Stoen R, Bergseng H, Flottorp ST, Mageroy G, Grunewaldt KH, Aker K. Immediate Skin-to-Skin Contact in Very Preterm Neonates and Early Childhood Neurodevelopment: A Randomized Clinical Trial. JAMA Netw Open. 2025 Apr 1;8(4):e255467. doi: 10.1001/jamanetworkopen.2025.5467. PMID 40238094
- [Derived] Kristoffersen L, Bergseng H, Engesland H, Bagstevold A, Aker K, Stoen R. Skin-to-skin contact in the delivery room for very preterm infants: a randomised clinical trial. BMJ Paediatr Open. 2023 Mar;7(1):e001831. doi: 10.1136/bmjpo-2022-001831. PMID 36958792